CLINICAL TRIAL: NCT03352791
Title: A Cluster Randomized Controlled Trial (RCT) of the Dementia Symptom Management (DSM) at Home Program Hospice Edition
Brief Title: The Dementia Symptom Management at Home Program Hospice Edition
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to operational changes at the participating agency.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 17-01080
Record Dates: First submitted 2017-11-21; First posted 2017-11-24 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DSM-H Hospice Edition (Active Comparator): training, assigning of champions to serve as mentors and performance improvement leads, and workflow changes including caregiver education pamphlets, interdisciplinary care plans, treatment algorithms, and assessment instruments.
  Interventions: Behavioral: DSM-H Hospice Edition performance improvement program
- Control Arm (Active Comparator): Usual Care
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: DSM-H Hospice Edition performance improvement program — Patients in the performance improvement group will receive care from a care team who has received the DSM-H Hospice Edition performance improvement program
  Arms: DSM-H Hospice Edition
Behavioral: Usual Care — control will receive usual care from a care team who has not received the performance improvement program.
  Arms: Control Arm

SUMMARY:
Alzheimer's Disease and Related Disorders (dementia) poses a significant challenge to our public health. While many persons with dementia are cared for by friends and family in the community with the assistance of home healthcare and hospice, most clinicians and agencies are ill prepared to care for this population and therefore have difficulty assisting patients and caregivers in maintaining quality of life leading to adverse patient outcomes, increased caregiver stress and burnout, and healthcare utilization. This study will utilize a cluster randomized controlled design with 6 care teams at a single study site to examine the ability of a multi-component evidence-based practice hospice care quality improvement program for registered nurses, social workers and chaplains to improve the quality of life and reduce healthcare utilization for persons with dementia and their informal caregiver.

ELIGIBILITY:
Inclusion Criteria:

* PWD over the age of 65
* Admitted to MJHS hospice agency
* The patient and family caregiver speak English and/or Spanish.
* The informal caregiver is ≥18 years of age and spends at least 8 hours per week with the patient.
* Patients who score ≥6 on the Quick Dementia Rating Scale (at least mild impairment).

Exclusion Criteria:

* Patients with a separate Axis 1 diagnosis other than forms of dementia, depression or anxiety.
* PWD residing in assisted living facilities, nursing homes or board and care homes
* PWD solely receiving infusion or home health aide services.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

PRIMARY OUTCOMES:
Reduction in pain (PAINAD) | Day 0 and Day 30
  pain assessment tool for use in persons with moderate to severe dementia who cannot provide reliable report, and will be used if the QDRS>12
Reduction in Behavioral and Psychological Symptoms of Dementia (BPSD) using Neuropsychiatric Inventory Questionnaire (NPI-Q): | Day 0 and Day 30
  13-item tool that measures caregiver perception of BPSD presence and severity in PWD

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Brody, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States